CLINICAL TRIAL: NCT05960448
Title: Autonomic Effects of Transcutaneous Spinal Cord Stimulation in Veterans With Spinal Cord Injury (SCI)
Brief Title: Autonomic Effects of Spinal Cord Stimulation in Spinal Cord Injury
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: James J. Peters Veterans Affairs Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Jill M. Wecht, Ed.D., Principal Investigator, James J. Peters Veterans Affairs Medical Center
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 1727500
Record Dates: First submitted 2023-07-17; First posted 2023-07-25 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: Orthostatic Hypotension
Keywords: neuromodulation; stimulation; exercise; hand bike; thermoregulation; cold room
MeSH Terms: conditions — Hypotension, Orthostatic; Motor Activity

STUDY DESIGN:
Who Masked: Participant
Masking Description: The participant will not know whether or not they are receiving spinal stimulation at any given session
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Transcutaneous Spinal Cord Stimulation (Experimental): The transcutaneous spinal cord stimulation used in this experiment is specific to each participant as determined in a previous study. Possible parameters include biphasic or monophasic, Russian or Nonrussian, a variety of pulse widths, and location of stimulation (T7-8, T9-10,- T11-12, L1-2). The amplitude of the stimulation also depends on the results of the mapping study. This stimulation will be delivered 30 minutes at a time.
  Interventions: Other: Transcutaneous Spinal Cord Stimulation (TSCS)
- Sham Transcutaneous Spinal Cord Stimulation (Sham Comparator): The sham stimulation will follow the above parameters but will only be delivered for a minute rather than the full 30 minutes.
  Interventions: Other: Sham Transcutaneous Spinal Cord Stimulation

INTERVENTIONS:
Other: Transcutaneous Spinal Cord Stimulation (TSCS) — This is electrical stimulation delivered to the spinal cord through the skin and tissue using a cathode electrode to deliver the stimulation and anode electrodes to ground the circuit.
  Other Names: transcutaneous spinal stimulation (TSS)
  Arms: Transcutaneous Spinal Cord Stimulation
Other: Sham Transcutaneous Spinal Cord Stimulation — This is designed to appear like transcutaneous spinal cord stimulation without actually delivering the stimulation.
  Other Names: Sham Transcutaneous Spinal Stimulation; Placebo Transcutaneous Spinal Stimulation; Placebo Transcutaneous Spinal Cord Stimulation
  Arms: Sham Transcutaneous Spinal Cord Stimulation

SUMMARY:
The goal of this interventional crossover study is to determine the effects of transcutaneous spinal cord stimulation (TSCS) on the ability to perform moderate exercise and regulate core body temperature in the chronic spinal cord injury community. The main questions it aims to answer are:

* What are the effects of active TSCS targeted for BP control on exercise endurance time and HR recovery during submaximal arm cycle ergometry (ACE) as compared to sham TSCS in participants with chronic, cervical SCI?
* What are the effects of active TSCS on Tcore responses to cool ambient exposure and on subjective reporting of thermal comfort and thermal sensitivity as compared to sham TSCS.

Participants will receive sham and active stimulation while using an arm bicycle or while in a cold room. Participants are free to participate in either the exercise phase, the cold room phase, or both phases of this study.

Please note that there no expected long term benefits of this study.

DETAILED DESCRIPTION:
The purpose of the first part of this research study is to determine the effects of active transcutaneous spinal cord stimulation (TSCS) targeted for blood pressure (BP) control on exercise endurance time and heart rate (HR) recovery time during an arm cycle test. The results will help guide experimental studies aimed at improving exercise, rehabilitation, health, and longevity in the SCI population. If the participant chooses to participate in part one of this study, the participant will be asked to visit the laboratory for 2 visits that take about 3-4 hours each.

The purpose of part two of this study is to compare the effects of electricity being delivered through surface electrodes (sticky pads on the participants skin), called active transcutaneous spinal cord stimulation (TSCS), compared to sham TSCS (sticky pads with electricity initially turned on but then turned off) on the participants ability to 1) keep the participants body temperature stable and 2) feel comfortable, while in a cool environment (cool room at 64° F) for 90 minutes. The investigators will assess the participant thermal sensation by asking the participant if overall they feel cold, cool, neutral, warm, or hot and their comfort level by asking the participant to grade their thermal comfort (how comfortable or how uncomfortable they feel) when the participant is seated in a thermoneutral room (80° F) and again in the cool room with active TSCS compared to the cool room with sham TSCS. The results will help guide experimental studies aimed at improving health and longevity in the population with SCI. If the participant chooses to participate in this study, there will be 2 study visits that last about 3-4 hours each.

ELIGIBILITY:
Inclusion Criteria:

* You are above the age of 18 years old
* You have an SCI between C3-T6
* You have been injured longer than 1 year
* You participated in a prior experiment "Targeted Transcutaneous Spinal Cord Stimulation to Restore Autonomic Cardiovascular Health in Individuals with Spinal Cord Injury"
* You have an American Spinal Injury Association injury classification scale (AIS) A, B, C
* Your prescription medications have not changed for at least 30 days

Exclusion Criteria:

* You have a history of seizures
* You have an acute illness or infection
* You have diabetes
* You have untreated thyroid disease
* You have a neurological condition other than SCI (Alzheimer's disease, dementia, stroke, multiple sclerosis, Parkinson's disease, etc.)
* You have a history of heart or vascular disease (coronary artery disease, congestive heart failure, peripheral artery disease,)
* You have a history of moderate or severe head trauma (TBI) or diagnosed with cognitive impairment
* You have a present or history of a psychological disorder
* You have contraindications to electricity over your spine
* You are dependent on a ventilator to breathe or have an open tracheostomy site
* You have a recent history of substance abuse (within the past 3 months)
* You have open wounds over the spine at the level targeted for stimulation
* You are pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-07-30 (Actual); Primary Completion 2026-07-30 (Estimated); Study Completion 2026-07-30 (Estimated)

PRIMARY OUTCOMES:
Exercise Endurance Time | During procedures (30 minutes)
  Total time (minutes) the participant is able to exercise during the submaximal arm cycle ergometry test.
Recovery Heart Rate | During procedures (60 minutes)
  Total time (minutes) for heart rate to return to baseline levels after submaximal exertion.
Tcore | During procedures (90 minutes)
  This outcome measure is measured in degrees Celsius.
Thermal Comfort | During procedures (90 minutes)
  Feeling of comfort from: +3 (very comfortable) to -3 (very uncomfortable).

SECONDARY OUTCOMES:
Workload | End of exercise (30 minutes)
  This outcome is measured in Watts (highest watt obtained)
Rate of Perceived Exhaustion | End of exercise (30 minutes)
  This is measured on the Borg scale (06-20) higher number = harder perceived exertion

CONTACTS AND LOCATIONS:
Overall Officials: Jill M Wecht, EdD, Principal Investigator — James J. Peters Veterans Affairs Medical Center
Locations (1):
- James J Peters VAMC, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: No